CLINICAL TRIAL: NCT00857454
Title: A Phase III Open-label Extension of the MTE08 Trial (A Phase III Open-label Titration Trial to Evaluate the Effectiveness and Safety of Different Doses of a Dermal Application of Testosterone MD-Lotion® (Cutaneous Solution) in Hypogonadal Men) to Evaluate Skin-safety
Brief Title: A Trial to Evaluate the Ongoing Skin Safety of Testosterone MD-Lotion Formulations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14273; MTE09 (Other: Acrux); I5E-MC-TSAI (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-03-04; First posted 2009-03-06 (Estimated); Results first posted 2011-01-05 (Estimated); Last update posted 2011-01-05 (Estimated); Status verified 2010-12

CONDITIONS: Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone Propionate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Testosterone MD-lotion (Experimental): In this open-label extension of the MTE08 trial, participants received Testosterone Metered Dose (MD)-Lotion for 60 days (dosing from Day 121 of the MTE08 trial to Day 180 of the MTE09 trial). Participants in MTE08 initially received 3.0 milliliters (mL) (60 micrograms [mg]) of 2% Testosterone MD-Lotion, and may have had their dose of testosterone adjusted upwards or downwards.
  Doses could be titrated to one of the following:
  1.5 mL (30 mg) of 2% Testosterone MD-Lotion applied daily by 2 doses to the axilla (1.5 mL to one axilla).
  3.0 mL (60 mg)of 2% Testosterone MD-Lotion applied daily by 2 doses to the axilla (1.5 mL to each axilla).
  4.5 mL (90 mg)of 2% Testosterone MD-Lotion applied daily by 3 doses to the axilla (2 x 1.5 mL to one axilla and 2 x 1.5 mL to the other axilla).
  6.0 (120 mg)of 2% Testosterone MD-Lotion applied daily by 4 doses to the axilla (2 x 1.5 mL to each axilla).
  Interventions: Drug: Testosterone MD-Lotion

INTERVENTIONS:
Drug: Testosterone MD-Lotion — 30 mg to 120 mg administered topically once daily for 60 days
  Other Names: LY900011; Axiron

SUMMARY:
Testosterone replacement treatment is the most effective way of treating hypogonadism in men. Acrux has a propriety testosterone replacement product, Testosterone MD-Lotion and this study will assess the occurrence of skin safety events for a further two months of continuous use of the Testosterone MD-Lotion® (cutaneous solution) after completion of the MTE08 (NCT00702650) trial.

ELIGIBILITY:
Inclusion Criteria:

* Hypogonadal males with a qualifying general medical health who have Completed the MTE08 trial up to and including Day 120/121 in a compliant manner
* Were able to communicate with the trial staff, understand the Trial Information Sheet and sign the Written Informed Consent Forms; were willing to follow the Protocol requirements and comply with Protocol restrictions and procedures

Exclusion Criteria:

* Any clinically significant chronic illness or finding and/or laboratory testing that would interfere with the trial objectives or safety of the subject
* Any man in whom testosterone therapy was contraindicated, which included those with:

  * Known or suspected carcinoma (or history of carcinoma) of the prostate or clinically significant symptoms of benign prostatic hyperplasia and/or clinically significant symptoms of lower urinary obstructions and with a International Prostate Symptoms Score (IPSS) score of greater than or equal to 19
  * Known or suspected carcinoma (or history of carcinoma) of the breast
  * Severe liver disease (i.e. cirrhosis, hepatitis or liver tumours or liver function tests >2 times the upper limit of the normal range values
  * Active deep vein thrombosis, thromboembolic disorders or a documented history of these conditions
  * Current significant cerebrovascular or coronary artery disease
  * Untreated sleep apnoea
  * Haematocrit of >54%
  * Untreated moderate to severe depression
* Men with clinically significant prostate exam or clinically significant elevated serum Prostate Specific Antigen (PSA) level (> 4 ng/mL) or age adjusted reference range of PSA values
* Men taking concomitant medications (prescribed, over-the-counter or complementary) that would affect Sex Hormone Binding Globulin (SHBG) or testosterone concentrations (excluding Testosterone MD-Lotion (cutaneous solution)) or metabolism such as warfarin, insulin, opiates, gonadotropin-releasing hormone analogues (GnRH), 5 alpha reductase inhibitors, propanolol, oxyphenbutazone, corticosteroids (except for physiological replacement doses), estradiol
* Men with uncontrolled diabetes (Hemoglobin A1c [HbA1c] greater than or equal to 10%)
* Subjects intending to have any surgical procedure during the course of the trial
* Subjects with a partner of child bearing potential who are not willing to use adequate contraception for the duration of the trial
* Subjects whose partners are pregnant

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- United States (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tuscon, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burbank, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Colorado Springs, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Britain, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ocala, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boise, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shawnee Mission, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label extension to the MTE08 trial. Only participants in the MTE08 trial who consented and met eligibility criteria could be enrolled in MTE09.
Pre-assignment Details: Participants received 3.0 mL (60 mg) of 2% Testosterone MD-Lotion for 60 days, and may have had their dose adjusted upwards or downwards (Subjects in MTE09 were continued on the dose that they were taking at the conclusion of study MTE08. A total of 2 patients received 30 mg; 49 remained on 60 mg, 12 received 90 mg; and 8 received 120 mg).
Groups:
- Testosterone MD-lotion: 30 to 120 mg of 2% Testosterone MD-Lotion administered topically once daily for 60 days
Period: Overall Study
Arm/Group | Testosterone MD-lotion
Started | 71
Completed | 51
Not Completed | 20
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 2
Not completed — Total Testosterone >1050 ng/dL | 1
Not completed — Total Testosterone <300 ng/dL | 8
Not completed — MTE09 enrollment criteria not met | 6

BASELINE CHARACTERISTICS:
Arm/Group | Testosterone MD-lotion
Number analyzed (Participants) | 71
Age Continuous [Mean (Standard Deviation); unit: years] | 52.3 (12.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 71
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 54
  African American | 6
  Hispanic | 10
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 71
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square metter (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms per square metter (kg/m^2) | 29.78 (3.61)
Baseline Total Testosterone Level [Mean (Standard Deviation); unit: nanograms per deciliter (ng/dL)] | 217.93 (84.70)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline MTE08 to MTE09 Endpoint in Draize Score
Description: Draize score is a measurement of skin irritability of the application site based on erythema/escar and oedema. Erythema/eschar scoring ranges from 0 (no erythema) to 4 (severe erythema [beet redness] to slight eschar formation [injuries in depth]). Oedema scoring ranges from 0 (no oedema) to 4 (severe oedema [raised more than 1 millimeter and extending beyond area of exposure]. The total Draize score ranges from 0 to 8.
Time Frame: Day 1, Day 190
Population: Participants enrolled in the study who had a baseline on MTE08 (Day 1) and a measurement at MTE09 endpoint (Day 190).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Testosterone MD-lotion
Number analyzed (Participants) | 68
units on a scale | 0.0 (0.12)

2. Secondary Outcome: Change From Baseline MTE08 to MTE09 Follow-up in Fasting Insulin
Time Frame: Day 1, up to Day 190
Population: Participants enrolled in the study who had a baseline on MTE08 (Day 1) and a measurement at endpoint (Day 180) or Follow-Up/Early Withdrawal (Day 190).
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Testosterone MD-lotion
Number analyzed (Participants) | 66
uIU/mL | 1.43 (11.23)

3. Secondary Outcome: Change From Baseline MTE08 to MTE09 Follow-up in Fasting Glucose
Time Frame: Day 1, up to Day 190
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Testosterone MD-lotion
Number analyzed (Participants) | 65
milligrams per deciliter (mg/dL) | 12.25 (35.56)

4. Secondary Outcome: Change From Baseline MTE08 to MTE09 Follow-up in Prostatic Specific Antigen (PSA)
Time Frame: Day 1, up to Day 190
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Testosterone MD-lotion
Number analyzed (Participants) | 67
nanograms per milliliter (ng/mL) | 0.10 (0.54)

5. Secondary Outcome: Change From Baseline MTE08 to MTE09 Follow-up in Luteinizing Hormone (LH) and Follicle Stimulating Hormone (FSH)
Time Frame: Day 1, up to Day 190
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Testosterone MD-lotion
Number analyzed (Participants) | 58
mIU/mL
  LH (N=50) | -1.39 (3.28)
  FSH (N=58) | -1.82 (3.87)

6. Secondary Outcome: Change From Baseline MTE08 to MTE09 Follow-up in Estradiol
Time Frame: Day 1, up to Day 190
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Testosterone MD-lotion
Number analyzed (Participants) | 32
picograms per milliliter (pg/mL) | 2.76 (18.97)

7. Secondary Outcome: Change From Baseline MTE08 to MTE09 Follow-up in Hemoglobin
Time Frame: Day 1, up to Day 190
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Testosterone MD-lotion
Number analyzed (Participants) | 67
grams per deciliter (g/dL) | 0.54 (1.160)

8. Secondary Outcome: Change From Baseline MTE08 to MTE09 Follow-up in Hematocrit
Time Frame: Day 1, up to Day 190
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of red blood cells in sample
Arm/Group | Testosterone MD-lotion
Number analyzed (Participants) | 66
percentage of red blood cells in sample | 0.03 (0.04)

ADVERSE EVENTS:
Arm/Group | Testosterone MD-lotion
Serious Adverse Events (participants affected / at risk) | 2/71
Other Adverse Events (participants affected / at risk) | 22/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone MD-lotion (N=71)
Hepatitis c (Infections and infestations) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone MD-lotion (N=71)
Cardiac flutter (Cardiac disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Application site erythema (General disorders) | 2 (2)
Application site irritation (General disorders) | 1 (1)
Application site oedema (General disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Peripheral coldness (General disorders) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Blood insulin increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Low density lipoprotein increased (Investigations) | 1 (1)
Prostatic specific antigen increased (Investigations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1)
Libido decreased (Psychiatric disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days